CLINICAL TRIAL: NCT01413360
Title: Phase 4 Study of High Dose Vitamin C in Chronic Hepatitis Patients
Brief Title: The Effect of High Dose Vitamin C on the Liver Function in Chronic Hepatitis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Hwan Yoon, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VitC
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Results first posted 2016-07-15 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Hepatitis; Chronic Hepatitis C; Chronic Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Chronic; Hepatitis C, Chronic; Hepatitis, Alcoholic | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HD Vitamin C (Experimental): High dose vitamin C
  Interventions: Drug: High dose vitamin C

INTERVENTIONS:
Drug: High dose vitamin C — Vitamin C, 3g per day (tid), with meal, per oral with water 100mL
  Other Names: Koreaeundan Vitamin C 1000

SUMMARY:
The investigators will evaluate the efficacy of high dose vitamin C in chronic hepatitis patients whose serum liver enzymes are elevated more than upper limit.

DETAILED DESCRIPTION:
The changes of laboratory findings including serum transaminase levels, serum albumin levels, Child-Pugh score, MELD score, and APRI score will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic hepatitis C patients

   * positive anti-HCV antibody more than 6 months
   * serum alanine aminotransferase 40 - 80 IU/L for more than 6 months
   * not indicated for antiviral therapy with interferon and ribavirin
2. Chronic alcoholic hepatitis

   * significant alcohol drinking history and no other cause of chronic hepatitis
   * serum alanine aminotransferase 40 - 80 IU/L for more than 6 months

Exclusion Criteria:

* Chronic hepatitis B, autoimmune hepatitis, primary biliary cirrhosis, Wilson's disease, hemochromatosis, other chronic hepatitis except chronic hepatitis C or alcoholic hepatitis
* decompensated liver cirrhosis
* platelet < 50,000/uL or white blood cell < 1,500/uL
* need and willing for antiviral therapy
* significant renal dysfunction (GFR < 30 mL/min/kg) or history of renal stone
* hepatotonic drug (i.e. silymarin, garlic oil, aronamin gold) usage within 2 weeks
* pregnancy, lactating woman

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Hwan Yoon, M.D, Ph.D, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HD Vitamin C
Started | 10
Completed | 7
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | HD Vitamin C
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 62 [39 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 10
Etiology [Number; unit: participants]
  HCV | 7
  Alcohol | 3
ALT [Median (Full Range); unit: IU/L] | 65 [41 to 142]

OUTCOME MEASURES:

1. Primary Outcome: The Change in Serum Alanine Aminotransferase Level From Baseline to 12 Weeks
Description: Serum alanine aminotransferase (ALT) level after 12 weeks of high dose vitamin C administration and Baseline serum ALT level
Time Frame: Baseline and 12 weeks
Measure: Median (Full Range); unit: IU/L
Arm/Group | HD Vitamin C
Number analyzed (Participants) | 7
IU/L
  ALT baseline | 77.5 [41 to 142]
  ALT 12 weeks | 105.5 [13 to 170]

2. Secondary Outcome: The Change in Serum Interleukin 22 Level From Baseline to 12 Weeks
Description: Serum interleukin 22(IL-22)level after 12 weeks of high vitamin C administration and Baseline IL-22 level
Time Frame: Baseline and 12 weeks
Measure: Median (Full Range); unit: pg/mL
Arm/Group | HD Vitamin C
Number analyzed (Participants) | 7
pg/mL
  IL-22 baseline | 3.66 [1.32 to 11.84]
  IL-22 after 12 weeks | 4.04 [0.32 to 5.2]

ADVERSE EVENTS:
Arm/Group | HD Vitamin C
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HD Vitamin C (N=10)
Dyspepsia (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No